CLINICAL TRIAL: NCT00482469
Title: The DIEP-Flap as a Model of Ischemia-Reperfusion
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Dr. R. van der Hulst, M.D., University Hospital Maastricht
Other Study IDs: MEC 07-2-004
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Ischemia-Reperfusion
Keywords: ischemia-reperfusion; ischemia; reperfusion; DIEP-flap; flap
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen tissue.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It is our goal to study the mechanism of ischemia-reperfusion injury. Our DIEP-operation is actually a clinical model of ischemia-reperfusion. Ischemia-reperfusion injury has never been directly studied in a human, clinical model of autologous transplant.

ELIGIBILITY:
Inclusion Criteria:

* patient is undergoing a DIEP-breast reconstruction, unilateral as well as bilateral
* is aged 18 years or older

Exclusion Criteria:

* diabetes mellitus
* diseases of the kidneys
* diseases of the liver
* patients who are taking immunosuppressants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical patients hospitalized for surgery.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-04; Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: René R Van der Hulst, MD, PhD, Study Chair — Maastricht University Hospital; Marieke GW Van den Heuvel, MD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Department of Plastic and Reconstructive surgery, Maastricht University Hospital, Maastricht, Netherlands

REFERENCES:
- [Derived] van den Heuvel MG, Bast A, Haenen GR, Ambergen AW, Mermans JF, van der Hulst RR. The role of antioxidants in ischaemia-reperfusion in a human DIEP flap model. J Plast Reconstr Aesthet Surg. 2012 Dec;65(12):1706-11. doi: 10.1016/j.bjps.2012.06.010. Epub 2012 Jul 11. PMID 22789619
- [Derived] van den Heuvel MG, Mermans JF, Ambergen AW, van der Hulst RR. Perfusion of the deep inferior epigastric perforator flap measured by laser Doppler imager. Ann Plast Surg. 2011 Jun;66(6):648-53. doi: 10.1097/SAP.0b013e3181e37bc8. PMID 21233705